CLINICAL TRIAL: NCT05944302
Title: Effect of Eye Movement Desensitization and Reprocessing (EMDR) on Pain in Patients With in Patients Rheumatoid Arthritis
Brief Title: EMDR on Pain in Patients With in Patients Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, müjde moran, head nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MesinU
Record Dates: First submitted 2023-06-09; First posted 2023-07-13 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Therapeutics
Keywords: Pain; EMDR; Patient; Rheumatoid Arthritis
MeSH Terms: conditions — Pain; Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: This study is two-stage. In the first stage, a randomized controlled trial type will be used to compare the effect of EMDR on pain in patients in the intervention and control groups, and in the second stage, a qualitative (qualitative) descriptive research type will be used to evaluate the experiences of the patients in the intervention group with the EMDR program.
Masking Description: In the study, block randomization will be done to eliminate selection bias and to provide balance in the number of individuals between groups. In this method, the number of groups and probabilities must be equal in each block. If we evaluate a study in which 2 different treatment methods (A and B) will be applied and the evaluations are equally probable; A total of 4 individuals are assigned to each block, with 2 subjects assigned to each treatment group. Thus, at the end of each quadruple assignment, the number of subjects in the 2 treatment groups is equalized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (EMDR) (Experimental): Since the aim of the study was to examine the effect of EMDR on pain, the pain levels of 32 the patients in the intervention group were examined before the first session and after the last session EMDR application. The control measurement was made 1 month after the last session of EMDR. To the initiative group; The first EMDR session was applied after the Personal Information Form and VAS were applied.
  The "Personal Information Form" was applied only once before the first session. Each EMDR session lasts between 45 and 90 minutes. EMDR was applied to the patients between 3-12 sessions. After the last EMDR session, "VAS" and "Individual In-depth Interview Question Form ". were applied.
  Interventions: Behavioral: EMDR group
- Control group (No Intervention): Pre-test (VAS) and post-test (VAS), and 1 month later, control measurement (VAS) data collection forms were applied simultaneously with the admitted 32 the patients. No application was made to the patients except for routine follow-up, anamnesis and medical treatment.

INTERVENTIONS:
Behavioral: EMDR group — Eye Movement Desensitization and Reprocessing
  Arms: Intervention group (EMDR)

SUMMARY:
They explained the improvement of pain in patients with EMDR treatment in chronic pain with Shapiro's adaptive information processing model. According to this model; The nociceptive sense is related to the emotional response. During the traumatic event, the painful stimulus is stored both physically and as an image, thought, and affect. Therefore, traumatic memories contain affective elements as well as conscious awareness and contribute significantly to stress along with chronic pain. Reprocessing these dysfunctionally stored memories will allow the problematic memories to integrate, resulting in both symptom relief and increased personal efficacy. According to the explanations made with the adaptive information processing model, the perception of the traumatic event is reprocessed with bidirectional stimulation given its somatic and affective components, and the cortical integration of the memory is provided. Changing the emotional dimension of pain may lead to changes in pain pathways, altering the memory and reproduction of pain in the nervous system. When desensitization is achieved against negative emotions; It has been hypothesized that once the patient has a more normal response to pain or stress, it will not revert to a limbic magnified response of pain unless a new trauma has been experienced. Painful conditions can continue to bother even after the illness or injury has been successfully treated. This may be the result of improperly stored memories and chronic active pain. In addition to medication, physical therapy, patient education and psychological support are very important in relieving rheumatological pain.

DETAILED DESCRIPTION:
In our study, it was considered to examine the effect of EMDR in reducing pain, one of the most common complaints of RA patients. Over time, the emotional discomfort caused by the pain increases with the persistence of the pain, and as a result, a medical condition causes a psychological problem to develop. Pain is a learned emotional experience. Therefore, psychological components should not be ignored in the evaluation of pain. At the end of EMDR sessions, patients are confident that they can effectively live with it, even if they have a very small amount of pain. He has learned to deal with pain without fear or anxiety. No more pain for the patient; It has become meaning "just an experience", realizing that living with pain is like traveling on a long road full of hidden pitfalls.

EMDR applications have been used in many treatment applications in recent years. The reasons for this are the rapid results after the treatment and the simplicity of the procedure. EMDR has been accepted as an evidence-based treatment method by the UK Department of Health (2001), the American Psychiatric Association (2004), the Australian Post Traumatic Mental Health Center (2007) and the Dutch National Mental Health Guidelines Guidance Committee (2003). The increasing prevalence of EMDR treatment in psychiatric nursing practice is based on the increasing number of scientifically based reports.

Studies have reported that EMDR application has positive effects on pain in different sample groups. In the literature review, it was seen that EMDR was applied to RA patients in only one study. In the study, 75 RA patients were divided into 2 intervention groups and a control group to compare the effect of EMDR and directed imagery on pain severity in RA patients. Between the two methods, it was concluded that EMDR was more effective on pain compared to the directed imagery and control group. It is assumed that EMDR can achieve beneficial results in RA patients.

The aim of the nursing approach is to enable the patient to recognize their psychological state, try to reduce their negative emotions and use coping methods.The nurse has the responsibility of educating patients about treatments, providing patient counseling, and supporting the patient to make informed decisions and take responsibility for self-care. He also needs to research about treatment options and follow up on current treatments and interventions. Considering all these factors, it is thought that EMDR, which will be applied to RA patients by specialist psychiatric nurses trained in this subject, can be used as an independent nursing practice in reducing pain and improving vital signs.

With this study the investigators planned, EMDR will be applied to RA patients, and it will be ensured that the data on whether this method is effective for pain will be brought to the literature. With the qualitative dimension, which is the second dimension of this study, which the investigators will bring to the literature, it will be ensured that the patients also express their feelings. In addition, this study will lead to the planning of new studies and publications, will reduce pain in patients with RA in whom EMDR is applied, will offer alternative options that specialist psychiatric nurses can apply in patients with pain, and will be a guiding resource for investigating the effect of EMDR on the pain of RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Under 18 years of age,
* Receiving another psychosocial therapy on working dates,
* Those who do not agree to participate in the research,
* Pregnancy,
* VAS pain score less than 4,
* Using analgesic medication at least 4 hours ago,
* Having a physical/mental disability or disability and illness that would prevent them from participating in EMDR,

Exclusion Criteria:

* Who cannot complete the EMDR application for any reason (health problem, not being able to spare time)
* Patients who want to leave the study voluntarily will be excluded from the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
visual analog scale (vas) | 1 year
  When patients talk about the event they experienced about their pain, they no longer feel discomfort, they learn to cope with their pain without fear or anxiety. It will result in them expressing that it has become "just a living experience" or completion. The scale consists of a 10 cm ruler on which there is no pain on one end and excruciating pain on the other end, on which the patient marks the pain. 1 indicates at least 10 most pain.

SECONDARY OUTCOMES:
Personal Information Form | 1 year
  This form, which was prepared by the researcher and developed by scanning the literature, consists of 14 questions. The personal information form consists of questions questioning sociodemographic characteristics (age, gender, marital status, etc.) and clinical characteristics (presence of chronic disease or pain, use of painkillers, etc.).

OTHER OUTCOMES:
Individual In-depth Interview Question Form | 1 year
  The Individual In-depth Interview Question Form created by the researcher in order to evaluate the experiences of RA patients with the EMDR program consists of 10 questions. The questionnaire was sent to five faculty members who are experts in the field of mental health and psychiatric nursing and expert opinion was obtained.There are no right or wrong answers to the questions. Questions do not have minimum and maximum values. These are qualitative questions to measure the experience of patients.

CONTACTS AND LOCATIONS:
Overall Officials: serpil yılmaz, Study Director — Mersin University; mualla yılmaz, Study Director — Mersin University
Locations (2):
- Turkey (Türkiye) (2):
  - Mersin University Hospital, Mersin, Yenişehir
  - Mersin University, Mersin, Yenişehir

IPD SHARING:
Plan to Share IPD: No
Effect of Eye Movement Desensitization and Reprocessing (EMDR) on Pain in Patients with in Patients Rheumatoid Arthritis

REFERENCES:
- See also: EMDR (With Eye Movements) Desensitization and Reconstruction Processing): Different in Psychotherapy One Option — https://dusunenadamdergisi.org/storage/upload/pdfs/1586350339-tr.pdf
- See also: Shapiro, F. (2001). Eye movement desensitization and reprocessing: Basic principles, proto — https://smartlib.umri.ac.id/assets/uploads/files/6cfb4-eye_movement_desensitization_and_reprocessing__emdr___basic_principles__protocols__and_procedures__2nd_edition.pdf
- See also: Sinici, E. (2016). Evaluation of EMDR therapy efficacy in the treatment of phantom pain. The Journal of Psychiatry and Neurological Sciences, 29:349-358 DOI: 10.5350/DAJPN2016290406 — https://arsiv.dusunenadamdergisi.org/tr/DergiPdf/DUSUNEN_ADAM_DERGISI_6eb40367c65a4a88af25e3aca7b8eac3.pdf

DOCUMENTS (1):
  • Informed Consent Form (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT05944302/ICF_000.pdf